CLINICAL TRIAL: NCT01708850
Title: A Pilot Study in Cancer Patients With Central Venous Catheter Associated Deep Vein Thrombosis in the Upper Extremity Treated With Rivaroxaban (Catheter 2)
Brief Title: Study in Cancer Patients With Central Line Associated Clots in the Upper Extremity Treated With Rivaroxaban (Catheter 2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Gwynivere Davies, Resident Researcher (Principal Investigator: Dr. Michael Kovacs, London Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Catheter 2
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Neoplasm; Central Venous Catheter Thrombosis
MeSH Terms: conditions — Neoplasms; Upper Extremity Deep Vein Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rivaroxaban (Other): Rivaroxaban 15 mg po bid x 3 weeks, followed by rivaroxaban 20 mg po daily x 9 weeks. Then up to discretion of investigator to decide regarding further anticoagulation as study length is limited to 12 weeks.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — All specified in arm description. One arm study.
  Other Names: Xarelto

SUMMARY:
Patients with cancer and an upper extremity DVT associated with a central venous catheter (CVC) will receive rivaroxaban. CVC survival will be assessed and compared to previous rates with low molecular weight heparin (LMWH) and warfarin, along with secondary safety outcomes including bleeding and recurrent venous thromboembolism.

The investigators hypothesize that anticoagulation with rivaroxaban in patients with UEDVT secondary to central venous catheters in patients with active malignancy is an effective therapy as quantified by the success of catheter preservation. Prolonged line salvage rate without recurrence of UEDVT will improve the management of cancer patients who develop an upper extremity deep venous thrombosis in the setting of a central venous catheter.

DETAILED DESCRIPTION:
This will be a prospective cohort study of patients who present with an acute upper limb thrombosis in the setting of a central venous catheter. The total study duration will be 12 weeks, with one follow up telephone visit at 6 months. All patients will be treated with rivaroxaban at a dose of 15 mg orally twice daily for three weeks, followed by 20 mg daily. Anticoagulation will continue for three months regardless of the length of time the catheter is in place. Continuation of anticoagulation beyond this time period is at the discretion of the investigators.

Strengths of this study include its prospective cohort format, and access to a large oncologic population through the London Regional Cancer Program and other corresponding centres. In addition, The Catheter Study looking at CVC survival and safety in patients with cancer diagnosed with UEDVT and treated with a bridging protocol of warfarin/dalteparin was organized primarily through the LHSc and results therein could be directly compared to the results from this study given the similar patient population.

Limitations of this study include the small sample size and the fact that there is no LMWH monotherapy comparison group. In addition, this will be an open study with no blinding, given the nature of line survival. There is also the chance that a proportion of patients will have their catheters removed for other reasons, such as finishing treatment or personal preference, which could affect the validity of survival results.

This design was selected given the small number of patients presenting with this diagnosis each year at our centre, which would present difficulty in accruing enough patients for several comparisons group. Results will be compared to the Catheter Study and previous literature.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age.
2. Symptomatic acute upper limb thrombosis in the axillary, subclavian, innominate or internal jugular veins, with or without pulmonary embolism, associated with central venous catheter objectively documented by compression ultrasonography, venogram or CT scan.
3. Diagnosis of active malignancy (other than non-melanoma skin cancer), defined as patients who are either receiving active treatment, or have metastatic disease or who have been diagnosed within the past two years.
4. Willing to provide written informed consent.

Exclusion Criteria:

1. Dialysis catheters.
2. Active bleeding or high risk for major bleeding.
3. Platelet Count < 75 x 109/L.
4. Creatinine Clearance < 30 mL/min.
5. Currently on other anticoagulant with therapeutic intent for another indication.*
6. Pulmonary embolism accompanied by hemodynamic instability or oxygen requirement.
7. Inability to infuse through the catheter after a trial of intraluminal thrombolytic therapy (ie. 2 mg tPA).
8. Patients with AML, ALL or multiple myeloma with a bone marrow or stem cell transplant planned within the next 3 months.
9. Thrombosis involving the brachial or cephalic veins only.
10. Treatment for current episode > 7 days with any acceptable anticoagulant therapy.
11. Concomitant use of P-glycoprotein and CYP3A4 inhibitors (ie. azole antifungals such as ketoconazole) or inducers (ie. rifampicin, antiepileptics).*
12. Recent coronary artery stent requiring dual anti-platelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-11; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of central line failure, defined as infusion failure that does not respond to 2mg tPA. | 12 weeks
  The primary endpoint of the study will be proportion of central line failure, defined as infusion failure that does not respond to 2mg tPA, within the 3 months of study follow-up.

SECONDARY OUTCOMES:
Recurrence of DVT or PE | 12 weeks
Major Bleeding | 12 weeks
Clinically Relevant Non-Major Bleeding | 12 weeks
Death | 12 weeks
Time to Central Line Failure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael J. Kovacs, MD, FRCPC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Kovacs MJ, Kahn SR, Rodger M, Anderson DR, Andreou R, Mangel JE, Morrow B, Clement AM, Wells PS. A pilot study of central venous catheter survival in cancer patients using low-molecular-weight heparin (dalteparin) and warfarin without catheter removal for the treatment of upper extremity deep vein thrombosis (The Catheter Study). J Thromb Haemost. 2007 Aug;5(8):1650-3. doi: 10.1111/j.1538-7836.2007.02613.x. Epub 2007 May 7. PMID 17488349